CLINICAL TRIAL: NCT05189665
Title: A Randomized Controlled Study on the Anatomical Reduction and Functional Recovery Effects of Two Transvaginal Apical Slings on Pelvic Organ Prolapse
Brief Title: the Anatomical Reduction and Functional Recovery Effects of Two Transvaginal Apical Slings on Pelvic Organ Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Sun Xiuli, Chief Gynecology Physician, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pkuh4
Record Dates: First submitted 2021-11-23; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-10

CONDITIONS: Pelvic Organ Prolapse
Keywords: Extraperitoneal high uterosacral ligament suspension
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extraperitoneal high sacral ligament suspension Group (Experimental): We will recruit 62 POP patients ,and perform Surgery Extraperitoneal high sacral ligament suspension surgery on them.
  Interventions: Procedure: Extraperitoneal high sacral ligament suspension surgery
- Sacrospinous Ligament Suspension Group (Active Comparator): We will recruit 62 POP patients ,and perform sacrospinous ligament suspension surgery on them.
  Interventions: Procedure: Sacrospinous ligament fixation

INTERVENTIONS:
Procedure: Extraperitoneal high sacral ligament suspension surgery — The extraperitoneal high sacral ligament suspension surgery is to shorten the bilateral uterosacral ligaments .
  Arms: Extraperitoneal high sacral ligament suspension Group
Procedure: Sacrospinous ligament fixation — The sacrospinous ligament fixation surgery is to open the front and back peritoneum through the vagina and shorten the bilateral uterosacral ligaments.
  Arms: Sacrospinous Ligament Suspension Group

SUMMARY:
The study is a prospective study at a single institution. Investigators create strict inclusion and exclusion criteria, selecting 124 patients with POP(≥II degree and have symptoms that need operation) . 62 patients in the intervention group accept extraperitoneal high uterosacral ligament suspension. The other 62 patients in the other group accept sacrospinous ligament suspension.

DETAILED DESCRIPTION:
Investigators evaluate all women's operation method, operation time, bleed volume, overactive bladder questionnaire, PFDI-20，ICIQ-SF, I-QoL, PISQ-12, PFIQ-7, UDI-6, pre- and post-operation (at 1 month, 3 months, 6months and 1 year).

ELIGIBILITY:
Inclusion Criteria:

Age ≥30 years old;

pelvic organ prolapse, with or without abnormal urination or defecation or sexual disturbance, which affects the quality of life

Pelvic organ prolapse quantitation (POP-Q) is greater than or equal to Those who are in stage II and have symptoms and require surgery

The patient agrees to conduct the study and can be followed up on time.

Exclusion Criteria:

Those who cannot tolerate surgery and anesthesia

Those who need to remove the uterus

Those who have removed the uterus

Those who cannot be followed up on time.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
changes in POP-Q score at different time nodes | pre-operation and post-operation(at 1month, 3 month, 6 month and a year)
  Gynecological examination

SECONDARY OUTCOMES:
UDI-6 scores at different time nodes UDI-6 | pre-operation and post-operation(at 1month, 3 month, 6 month and a year)
  Questionnaires on lower urinary tract symptoms and quality of life
Postoperative urinary incontinence assessment | post-operation(at 1month, 3 month, 6 month and a year)
  One hour pad test
OABss score at different time nodes | post-operation(at 1month, 3 month, 6 month and a year)
  Questionnaires lower urinary tract symptoms
PFDI-20 score at different time nodes | post-operation(at 1month, 3 month, 6 month and a year)
  Questionnaires on pelvic floor function and lower urinary tract symptoms and quality of life
ICIQ-SF score at different time nodes | post-operation(at 1month, 3 month, 6 month and a year)
  Questionnaires on lower urinary tract symptoms
I-QoL score at different time nodes | post-operation(at 1month, 3 month, 6 month and a year)
  Questionnaires on lower urinary tract symptoms and quality of life
PISQ-12 score at different time nodes | post-operation(at 1month, 3 month, 6 month and a year)
  Questionnaires on pelvic floor function and lower urinary tract symptoms and sexual quality of life
PFIQ-7 score at different time nodes | post-operation(at 1month, 3 month, 6 month and a year)
  Questionnaires on pelvic floor function and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: xiuli sun, professor, Study Chair — Beijing Key Laboratory of Female Pelvic Floor Disorders
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Extraperitoneal high uterosacral ligament sling is effective in treating pelvic organ prolapse, and postoperative anatomical recovery is good, not inferior to traditional sacral ligament sling
Supporting Information: Study Protocol, CSR
Time Frame: 2 years